CLINICAL TRIAL: NCT01214915
Title: A Phase 3, Open-label, Single-arm Study Evaluating the Effect of SPD422 on Platelet Lowering and Safety in Japanese Adults With At Risk Essential Thrombocythaemia Who Are Intolerant or Refractory to Current Cytoreductive Treatment
Brief Title: Effect of SPD422 on Platelet Lowering and Safety in Japanese Adults With At Risk Essential Thrombocythaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD422-308
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Essential Thrombocythemia (ET)
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — anagrelide

ARMS (1):
- Anagrelide Hydrochloride (Experimental)
  Interventions: Drug: Anagrelide Hydrochloride

INTERVENTIONS:
Drug: Anagrelide Hydrochloride — Subjects will be started at 1.0 mg per day and titrated as necessary.
  Other Names: SPD422

SUMMARY:
The purpose of this study is to investigate how effective and safe SPD422 (Anagrelide Hydrochloride) is in Japanese subjects, diagnosed with Essential Thrombocythemia, who's previously treatment has either not been effective or has caused unacceptable adverse reactions. The study will aim to show that platelet counts can be safely reduced in treated patients to below 600 x 10^9/L after a minimum of three months treatment. To demonstrate an positive effect platelet levels will need to remain below 600 x 10^9/L for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have previously been treated with a cytoreductive therapy and been intolerant or refractory to that therapy.

Exclusion Criteria:

* Subjects should not have any other underlying conditions or medications that would confound the study analysis or interact with the study medication.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-10-27 (Actual); Primary Completion 2012-10-24 (Actual); Study Completion 2012-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- Japan (19):
  - Akita University Hospital, Akita, Akita
  - Juntendo University Hospital, Hongo 3-1-3, Bunkyo-ku
  - Tokyo Metropolitan Cancer and Infectious diseases Center Kom, Honkomagome 3-18-22, Bunkyo-ku
  - Nippon Medical School Hospital, Sendagi 1-1-5, Bunkyo-ku
  - Chiba University Hospital, Chuo-ku Inohana 1-8-1, Chiba-shi
  - NHO Nagoya Medical Center, Nagoya, Chubu
  - Hokkaido University Hospital, Sapporo, Hokkaidō Prefecture
  - Juntendo University Shizuoka Hospital, Nagaoka, Izunokuni-shi
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Osaka City University Hospital, Osaka, Kansai
  - Gunma University Hospital, Showa-machi 3-39-15, Maebashi-shi
  - NHO Tokyo Medical Center, Higashigaoka 2-5-1, Meguro-ku
  - Mie University Hospital, Tsu, Mie-ken
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Niigata Cancer Center Hospital, Chuo-ku Kawagishi-cho 2-15-3, Niigata-shi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka University Hospital, Suita-shi, Osaka
  - Tokushima University Hospital, Tokushima, Tokushima Perfecture
  - Keio University Hospital, Tokyo

REFERENCES:
- [Result] Kanakura Y, Miyakawa Y, Wilde P, Smith J, Achenbach H, Okamoto S. Phase III, single-arm study investigating the efficacy, safety, and tolerability of anagrelide as a second-line treatment in high-risk Japanese patients with essential thrombocythemia. Int J Hematol. 2014 Oct;100(4):353-60. doi: 10.1007/s12185-014-1631-x. Epub 2014 Aug 27. PMID 25160063

RESULTS

PARTICIPANT FLOW:
Groups:
- Anagrelide Hydrochloride: Subjects will be started at 1.0 mg per day orally and titrated as necessary.
Period: Overall Study
Arm/Group | Anagrelide Hydrochloride
Started | 53
Completed | 42
Not Completed | 11
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (13.1)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 12
  50 - 59 years | 5
  60 - 69 years | 18
  70 - 79 years | 17
  >= 80 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 23
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Responded in Platelet Count
Description: A response was defined as platelet counts to <600x10^9/L across consecutive visits for at least 4 weeks following at least 3 months of treatment.
Time Frame: 12 months
Population: Full Analysis Set defined as subjects who had taken at least 1 dose of study medication and had at least 1 post-baseline platelet measurement assessment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 53
percentage of subjects | 67.9 [53.7 to 80.1]

2. Secondary Outcome: Percentage of Subjects With at Least 50% Reduction in Platelet Count
Description: Subjects who achieved at least 50% reduction in platelet count from their baseline level across consecutive visits for at least 4 weeks and following 3 months of treatment.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 53
percentage of subjects | 50.9 [36.8 to 64.9]

3. Secondary Outcome: Percentage of Subjects With Normalization in Platelet Count
Description: Normalization was defined as platelet counts ≤400x10^9/L across consecutive visits for at least 4 weeks following at least 3 months of treatment.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 53
percentage of subjects | 45.3 [31.6 to 59.6]

4. Secondary Outcome: Percentage of Subjects Who Responded in Platelet Count Whose Baseline Platelet Count Was ≥600x10^9/L
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 47
percentage of subjects | 68.1 [52.9 to 80.9]

5. Secondary Outcome: Percentage of Subjects Who Responded in Platelet Count Whose Baseline Platelet Count Was <600x10^9/L
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 6
percentage of subjects | 66.7 [22.3 to 95.7]

ADVERSE EVENTS:
Arm/Group | Anagrelide Hydrochloride
Serious Adverse Events (participants affected / at risk) | 15/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anagrelide Hydrochloride (N=53)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
CYTOGENETIC ABNORMALITY (Congenital, familial and genetic disorders) | 2 (2)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1)
COLONIC POLYP (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1)
OEDEMA (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 1 (1)
ANGIOIMMUNOBLASTIC T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CEREBRAL INFARCTION (Vascular disorders) | 2 (2)
LACUNAR INFARCTION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anagrelide Hydrochloride (N=53)
ANAEMIA (Blood and lymphatic system disorders) | 25 (27)
EOSINOPHILIA (Blood and lymphatic system disorders) | 3 (3)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
PALPITATIONS (Cardiac disorders) | 20 (23)
VERTIGO (Ear and labyrinth disorders) | 4 (6)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 (5)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (6)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
DENTAL CARIES (Gastrointestinal disorders) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 17 (20)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 3 (4)
GASTRITIS (Gastrointestinal disorders) | 4 (8)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 7 (9)
NAUSEA (Gastrointestinal disorders) | 5 (5)
VOMITING (Gastrointestinal disorders) | 5 (6)
CHEST PAIN (General disorders) | 3 (4)
FATIGUE (General disorders) | 9 (12)
MALAISE (General disorders) | 4 (4)
OEDEMA (General disorders) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 14 (17)
PYREXIA (General disorders) | 9 (10)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 3 (3)
BRONCHITIS (Infections and infestations) | 3 (3)
CYSTITIS (Infections and infestations) | 3 (4)
GASTROENTERITIS (Infections and infestations) | 3 (3)
HERPES ZOSTER (Infections and infestations) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 12 (19)
PHARYNGITIS (Infections and infestations) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (7)
CONTUSION (Injury, poisoning and procedural complications) | 6 (7)
FALL (Injury, poisoning and procedural complications) | 4 (4)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (6)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 7 (8)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 3 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5)
HEADACHE (Nervous system disorders) | 24 (31)
HYPOAESTHESIA (Nervous system disorders) | 6 (8)
POLLAKIURIA (Renal and urinary disorders) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (8)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 4 (4)
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 4 (4)
HYPERTENSION (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.